CLINICAL TRIAL: NCT06430567
Title: Comparing the Effectiveness of Blood Flow Restriction Training and Traditional Resistance Training in Post-surgery Rehabilitation of Latarjet Procedure
Brief Title: Blood Flow Restriction in Post-surgery Rehabilitation of Latarjet Procedure
Acronym: BFR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ensemble Hospitalier de la Côte (Other)
Responsible Party: Principal Investigator, Arnaud Meylan, Doctor, Ensemble Hospitalier de la Côte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EHC Morges BFR
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Shoulder Dislocation
Keywords: Blood flow restriction; Latarjet surgery; Rehabilitation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants between placebo and intervention group will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Patient will not use BFR
- Placebo 10% of pressure for arterial occlusion (Placebo Comparator): Patient will use BFR sub optimally as described in the literature
  Interventions: Device: Blood flow restriction (10% AOP compression) in the rehabilitation phase after Latarjet surgery for chronic shoulder instability
- Interventional 50% of pressure for arterial occlusion (Experimental): Patient will use the minimal pressure of 50% of arterial occlusion known to be effective in the literature
  Interventions: Device: Blood flow restriction (50% AOP compression) in the rehabilitation phase after Latarjet surgery for chronic shoulder instability

INTERVENTIONS:
Device: Blood flow restriction (50% AOP compression) in the rehabilitation phase after Latarjet surgery for chronic shoulder instability — Participants undergoing shoulder instability surgery (Latarjet procedure) by a single surgeon will receive standard physiotherapy (2 sessions per week) before being randomized into 3 groups at their 6th postoperative week check-up:
  Group 1) BFR Group with 50% AOP compression
  Group 1 will perform a 30-minute strengthening session twice weekly during postoperative weeks 7 to 14. They will do 4 exercises, completing 4 sets with 30-second rest intervals and 1 minute between exercises, following 30-15-15-15 at 40% 1RM (repetition maximum)
  Exercise :
  External rotation with pulley/band Internal rotation with pulley/band Frontal elevation with hyperpronation Diagonal abduction-external rotation with pulley/band
  BFR training will use the MadUp© system, placing the band proximally on the operated arm, with a central unit continuously monitoring and calibrating arm pressure.
  Arms: Interventional 50% of pressure for arterial occlusion
Device: Blood flow restriction (10% AOP compression) in the rehabilitation phase after Latarjet surgery for chronic shoulder instability — Participants undergoing shoulder instability surgery (Latarjet procedure) by a single surgeon will receive standard physiotherapy (2 sessions per week) before being randomized into 3 groups at their 6th postoperative week check-up:
  Group 2) BFR Group with 10% AOP compression
  Group 2 will perform a 30-minute strengthening session twice weekly during postoperative weeks 7 to 14. They will do 4 exercises, completing 4 sets with 30-second rest intervals and 1 minute between exercises, following 15-15-15-15 at 70% 1RM
  Exercise :
  External rotation with pulley/band Internal rotation with pulley/band Frontal elevation with hyperpronation Diagonal abduction-external rotation with pulley/band
  BFR training will use the MadUp© system, placing the band proximally on the operated arm, with a central unit continuously monitoring and calibrating arm pressure.
  Arms: Placebo 10% of pressure for arterial occlusion

SUMMARY:
The goal of this clinical trial is to evaluate the effects of Blood Flow Restriction (BFR) training on post-surgery rehabilitation following the Latarjet procedure in athletes aged 18-35.

The main questions it aims to answer are:

Does BFR training improve scapular belt muscle strength post-surgery? Does BFR training enhance shoulder function during rehabilitation?

Researchers will compare three groups:

BFR Group with 50% AOP [arterial occlusion pressure] compression BFR Placebo Group with 10% AOP compression Control Group

Participants will:

Perform the same four strengthening exercises twice a week Complete 16 semi-autonomous strength training sessions over 8 weeks Undergo isokinetic and isometric strength tests, shoulder mobility assessments, and complete self-assessment questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years
* Indication for shoulder stabilization surgery using the Latarjet procedure (documented anterior dislocations with proof of emergency reduction, with or without hypermobility and confirmation of traumatic capsulo-ligamentous injury by MRI).
* Regular exercise (min. 1x / week)
* Signed the informed consent form for the study.

Exclusion Criteria:

* Pregnant or breast-feeding women
* Active oncological disease under treatment. (Patient with stable oncological disease eligible)
* Adverse events during the 6-week post-operative period such as:-Fracture/displacement of the reconstructed bone-Luxation of the operated shoulder-Requirement for emergency hospitalization
* History of deep vein thrombosis/pulmonary embolism
* Inability to follow study procedures, due to language problems, psychological disorders, dementia.
* Need for skin grafting following shoulder stabilization surgery
* Coronary heart disease
* Unstable hypertension
* Peripheral vascular disease
* Hypercoagulable states (blood coagulation disorders)
* Left ventricular dysfunction
* Hemophilia

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Isokinetic strength | Preoperative and at 14 weeks postoperative
  Concentric peak torque (Nm) IR-ER at 60°/sec
Isokinetic strength | Preoperative and at 14 weeks postoperative
  Concentric peak torque (Nm) IR-ER at 240°/sec
Isokinetic strength | Preoperative and at 14 weeks postoperative
  Eccentric peak torque (Nm) IR-ER at 60°/sec
Isokinetic strength | Preoperative and at 14 weeks postoperative
  Concentric ratio (ER conc 60°/ IR conc 60°)
Isokinetic strength | Preoperative and at 14 weeks postoperative
  Cocking gesture ratio (IR exc 60° /ER conc 240°)
Isometric strength | Preoperative and at 14 weeks postoperative
  Flexion in the scapular plane (Nm)
Isometric strength | Preoperative and at 14 weeks postoperative
  Athletic shoulder test (positions I, Y, T) (Nm)
Isometric strength | Preoperative and at 14 weeks postoperative
  Grip test (Nm)

SECONDARY OUTCOMES:
Shoulder mobility | Preoperative and at 14 weeks postoperative
  Flexion
Shoulder mobility | Preoperative and at 14 weeks postoperative
  Abduction
Shoulder mobility | Preoperative and at 14 weeks postoperative
  Internal rotation at 90° abduction
Shoulder mobility | Preoperative and at 14 weeks postoperative
  External rotation at 90° abduction
Shoulder mobility | Preoperative and at 14 weeks postoperative
  Scapular dyskinesis test (SDT)
Scapular girdle stability | Preoperative and at 14 weeks postoperative
  Modified closed kinetic upper extremity stability test
Scapular girdle stability | Preoperative and at 14 weeks postoperative
  Shoulder Instability Return to Sport Index (SIRSI)
Scapular girdle stability | Preoperative and at 14 weeks postoperative
  Western Ontario Shoulder Instability Index (WOSI)

CONTACTS AND LOCATIONS:
Overall Officials: Bauer Stefan, MD, Study Director — EHC Morges

IPD SHARING:
Plan to Share IPD: No